CLINICAL TRIAL: NCT00287729
Title: A Randomized, Double-Blind, Placebo Controlled, Phase 3 Study of the Safety and Efficacy of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Safety and Efficacy of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PIPF-006; Capacity 1
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2011-06-13 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic; Pulmonary; Fibrosis; Lung; Pirfenidone; InterMune
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2403 mg/day pirfenidone (Active Comparator): 2403 mg/day pirfenidone dose group.
  Interventions: Drug: Pirfenidone
- placebo (Placebo Comparator): Placebo equivalent.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone — 2403 mg/day given orally, and administered in divided doses three times daily with food, for the duration of the study.
  Arms: 2403 mg/day pirfenidone
Drug: Placebo — Placebo equivalent, given orally, and administered in divided doses three times daily with food, for the duration of the study.
  Arms: placebo

SUMMARY:
The purposes of this study are to assess the efficacy of treatment with pirfenidone 2403 milligrams per day compared with placebo in patients with idiopathic pulmonary fibrosis (IPF)and to assess the safety of treatment with pirfenidone 2403 milligrams per day compared with placebo in patients with idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, safety and efficacy study of pirfenidone in patients with idiopathic pulmonary fibrosis (IPF). Approximately 320 patients at approximately 50 centers will be randomly assigned (1:1) to receive pirfenidone 2403 milligrams or placebo equivalent administered in divided doses three times per day (TID) with food. The primary outcome variable will be the absolute change in percent predicted Forced Vital Capacity from Baseline to Week 72. Patients will be randomized by geographic region.

Patients will receive blinded study treatment from the time of randomization until the last patient randomized has been treated for 72 weeks. A Data Monitoring Committee (DMC) will periodically review safety and efficacy data to ensure patient safety.

After week 72, patients who meet the Progression of Disease (POD) definition, which is a ≥ 10% absolute decrease in percent predicted Forced Vital Capacity or a ≥ 15% absolute decrease in percent predicted carbon monoxide diffusing capacity (DLco), will be eligible to receive permitted idiopathic pulmonary fibrosis therapies in addition to their blinded study drug. Permitted idiopathic pulmonary therapies include corticosteroids, azathioprine, cyclophosphamide and N-acetyl-cysteine (with restrictions).

ELIGIBILITY:
Primary Inclusion criteria:

* diagnosis of idiopathic pulmonary fibrosis
* 40 to 80 years of age
* Forced Vital Capacity ≥ 50% predicted value
* carbon monoxide diffusing capacity (DLco) ≥ 35% predicted value
* either Forced Vital Capacity or carbon monoxide diffusing capacity (DLco) ≤ 90% predicted value
* no improvement in past year
* able to walk 150 meters in 6 minutes and maintain saturation ≥ 83% while on no more than 6 liters per minute supplemental oxygen

Primary Exclusion criteria:

* unable to undergo pulmonary function testing
* evidence of significant obstructive lung disease or airway hyper-responsiveness
* in the clinical opinion of the investigator, the patient is expected to need and be eligible for a lung transplant within 72 weeks of randomization
* active infection
* liver disease
* cancer or other medical condition likely to result in death within 2 years
* diabetes
* pregnancy or lactation
* substance abuse
* personal or family history of long QT syndrome
* other IPF treatment
* unable to take study medication
* withdrawal from other IPF trials

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2006-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- InterMune, Inc., Brisbane, California, United States

REFERENCES:
- [Derived] Behr J, Nathan SD, Costabel U, Albera C, Wuyts WA, Glassberg MK, Haller H Jr, Alvaro G, Gilberg F, Samara K, Lancaster L. Efficacy and Safety of Pirfenidone in Advanced Versus Non-Advanced Idiopathic Pulmonary Fibrosis: Post-Hoc Analysis of Six Clinical Studies. Adv Ther. 2023 Sep;40(9):3937-3955. doi: 10.1007/s12325-023-02565-3. Epub 2023 Jun 30. PMID 37391667
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625
- [Derived] Kreuter M, Lee JS, Tzouvelekis A, Oldham JM, Molyneaux PL, Weycker D, Atwood M, Kirchgaessler KU, Maher TM. Monocyte Count as a Prognostic Biomarker in Patients with Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med. 2021 Jul 1;204(1):74-81. doi: 10.1164/rccm.202003-0669OC. PMID 33434107
- [Derived] Glassberg MK, Nathan SD, Lin CY, Morgenthien EA, Stauffer JL, Chou W, Noble PW. Cardiovascular Risks, Bleeding Risks, and Clinical Events from 3 Phase III Trials of Pirfenidone in Patients with Idiopathic Pulmonary Fibrosis. Adv Ther. 2019 Oct;36(10):2910-2926. doi: 10.1007/s12325-019-01052-y. Epub 2019 Aug 10. PMID 31401786
- [Derived] Nathan SD, Costabel U, Albera C, Behr J, Wuyts WA, Kirchgaessler KU, Stauffer JL, Morgenthien E, Chou W, Limb SL, Noble PW. Pirfenidone in patients with idiopathic pulmonary fibrosis and more advanced lung function impairment. Respir Med. 2019 Jul;153:44-51. doi: 10.1016/j.rmed.2019.04.016. Epub 2019 Apr 24. PMID 31153107
- [Derived] Kreuter M, Lederer DJ, Molina-Molina M, Noth I, Valenzuela C, Frankenstein L, Weycker D, Atwood M, Kirchgaessler KU, Cottin V. Association of Angiotensin Modulators With the Course of Idiopathic Pulmonary Fibrosis. Chest. 2019 Oct;156(4):706-714. doi: 10.1016/j.chest.2019.04.015. Epub 2019 Apr 29. PMID 31047956
- [Derived] Nathan SD, Costabel U, Glaspole I, Glassberg MK, Lancaster LH, Lederer DJ, Pereira CA, Trzaskoma B, Morgenthien EA, Limb SL, Wells AU. Efficacy of Pirfenidone in the Context of Multiple Disease Progression Events in Patients With Idiopathic Pulmonary Fibrosis. Chest. 2019 Apr;155(4):712-719. doi: 10.1016/j.chest.2018.11.008. Epub 2018 Nov 22. PMID 30472023
- [Derived] Nathan SD, Lancaster LH, Albera C, Glassberg MK, Swigris JJ, Gilberg F, Kirchgaessler KU, Limb SL, Petzinger U, Noble PW. Dose modification and dose intensity during treatment with pirfenidone: analysis of pooled data from three multinational phase III trials. BMJ Open Respir Res. 2018 Aug 2;5(1):e000323. doi: 10.1136/bmjresp-2018-000323. eCollection 2018. PMID 30116539
- [Derived] Neighbors M, Cabanski CR, Ramalingam TR, Sheng XR, Tew GW, Gu C, Jia G, Peng K, Ray JM, Ley B, Wolters PJ, Collard HR, Arron JR. Prognostic and predictive biomarkers for patients with idiopathic pulmonary fibrosis treated with pirfenidone: post-hoc assessment of the CAPACITY and ASCEND trials. Lancet Respir Med. 2018 Aug;6(8):615-626. doi: 10.1016/S2213-2600(18)30185-1. Epub 2018 Jun 29. PMID 30072107
- [Derived] Paterniti MO, Bi Y, Rekic D, Wang Y, Karimi-Shah BA, Chowdhury BA. Acute Exacerbation and Decline in Forced Vital Capacity Are Associated with Increased Mortality in Idiopathic Pulmonary Fibrosis. Ann Am Thorac Soc. 2017 Sep;14(9):1395-1402. doi: 10.1513/AnnalsATS.201606-458OC. PMID 28388260
- [Derived] Kreuter M, Bonella F, Maher TM, Costabel U, Spagnolo P, Weycker D, Kirchgaessler KU, Kolb M. Effect of statins on disease-related outcomes in patients with idiopathic pulmonary fibrosis. Thorax. 2017 Feb;72(2):148-153. doi: 10.1136/thoraxjnl-2016-208819. Epub 2016 Oct 5. PMID 27708114
- [Derived] Nathan SD, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, Glasscock KF, King TE Jr, Lancaster L, Lederer DJ, Lin Z, Pereira CA, Swigris JJ, Valeyre D, Noble PW, Wells AU. Effect of continued treatment with pirfenidone following clinically meaningful declines in forced vital capacity: analysis of data from three phase 3 trials in patients with idiopathic pulmonary fibrosis. Thorax. 2016 May;71(5):429-35. doi: 10.1136/thoraxjnl-2015-207011. Epub 2016 Mar 11. PMID 26968970
- [Derived] Lancaster L, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, King TE Jr, Lederer DJ, Lin Z, Nathan SD, Pereira CA, Swigris JJ, Valeyre D, Noble PW. Safety of pirfenidone in patients with idiopathic pulmonary fibrosis: integrated analysis of cumulative data from 5 clinical trials. BMJ Open Respir Res. 2016 Jan 12;3(1):e000105. doi: 10.1136/bmjresp-2015-000105. eCollection 2016. PMID 26835133
- [Derived] Noble PW, Albera C, Bradford WZ, Costabel U, Glassberg MK, Kardatzke D, King TE Jr, Lancaster L, Sahn SA, Szwarcberg J, Valeyre D, du Bois RM; CAPACITY Study Group. Pirfenidone in patients with idiopathic pulmonary fibrosis (CAPACITY): two randomised trials. Lancet. 2011 May 21;377(9779):1760-9. doi: 10.1016/S0140-6736(11)60405-4. Epub 2011 May 13. PMID 21571362

RESULTS

PARTICIPANT FLOW:
Groups:
- Pirfenidone (2403 mg/d): pirfenidone, total daily dose of 2403 mg/day, given as 3 divided doses 3 times/day
- Placebo: placebo equivalent, given as 3 divided doses 3 times/day
Period: Overall Study
Arm/Group | Pirfenidone (2403 mg/d) | Placebo
Started | 171 | 173
Completed | 137 | 142
Not Completed | 34 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pirfenidone (2403 mg/d) | Placebo | Total
Number analyzed (Participants) | 171 | 173 | 344
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 61 | 131
  >=65 years | 101 | 112 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (7.90) | 67.0 (7.80) | 66.9 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 123 | 124 | 247
Region of Enrollment [Number; unit: participants]
  United States | 148 | 150 | 298
  Europe | 23 | 22 | 45
  Australia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Vital Capacity(FVC)
Description: Mean Change in Percent Predicted Forced Vital Capacity (FVC) as measured from baseline to week 72. It is calculated as the simple difference between baseline Percent Predicted FVC measurements and week 72 Percent Predicted FVC measurements.
Time Frame: Baseline to week 72
Population: A modified intent-to-treat population of all randomized patients who received any amount of study drug is the primary population for efficacy and safety analyses. Missing FVC data due to death were assigned the worst rank and missing FVC data due to reasons other than death were imputed using the SSD method.
Measure: Mean (Standard Deviation); unit: Change in Percent Predicted FVC
Arm/Group | Pirfenidone (2403 mg/d) | Placebo
Number analyzed (Participants) | 171 | 173
Change in Percent Predicted FVC | -9 (19.58) | -10 (19.12)

2. Secondary Outcome: Categorical Assessment of Absolute Change in Percent Predicted Forced Vital Capacity
Description: Based on the change in baseline percent predicted FVC at week 72, patients were assigned to 1 of 5 categories: mild decline (<10% but >=0% decline), moderate decline (<20% but >=10% decline), severe decline (>=20% decline), mild improvement (>0% but <10% improvement), or moderate improvement (>=10% improvement). Those who died or had a lung transplant before Week 72 were included in the severe decline category. The results indicate the number of patients who experience Categorical Change in Percent Predicted Forced Vital Capacity.
Time Frame: Baseline to week 72
Population: A modified intent-to-treat population of all randomized patients who received any amount of study drug is used as the primary population for all efficacy and safety analyses. Missing data were imputed by the SSD method if the patient was alive and imputed to 0% if the patient died before the protocol-specified time point.
Measure: Number; unit: Patients
Arm/Group | Pirfenidone (2403 mg/d) | Placebo
Number analyzed (Participants) | 171 | 173
Patients
  Decline >=20% or death or lung transplantation | 20 | 23
  Decline <20% but >= 10% | 19 | 23
  Decline <10% but > 0% | 88 | 89
  Improvement of >=0% but <10% | 41 | 33
  Improvement of >=10% | 3 | 5

3. Secondary Outcome: Progression-free Survival
Description: Progression is defined as the first occurrence of a 10% absolute decline from baseline in percent predicted Forced Vital Capacity, a 15% absolute decline from baseline in percent predicted hemoglobin(Hgb)-corrected carbon monoxide diffusing capacity (DLco), or, death.
Time Frame: Baseline to Week 72
Population: A modified intent-to-treat population of all randomized patients who received any amount of study drug is used as the primary population for efficacy and safety analyses.
Measure: Number; unit: Number of Patients with Progression
Arm/Group | Pirfenidone (2403 mg/d) | Placebo
Number analyzed (Participants) | 171 | 173
Number of Patients with Progression
  Death or Disease Progression | 54 | 60
  Decline in percent predicted FVC >=10% | 31 | 41
  Decline in percent predicted DLco >=15% | 10 | 9
  Death Before Disease Progression | 13 | 10

4. Secondary Outcome: Change in the Six-Minute Walk Test (6MWT) Distance
Description: The change from Baseline to week 72 in distance walked during the 6-Minute Walk Test. This measure was calculated as the simple difference between baseline distanced walked over 6 minutes and week 72 distance walked over 6 minutes as measured in meters (m).
Time Frame: Baseline to Week 72
Population: A modified intent-to-treat population of all randomized patients who received any amount of study drug is used as the primary population for efficacy and safety analyses. Missing data were imputed by the SSD method if the patient was alive and imputed to 0 meters if the patient had died before the protocol-specified time point.
Measure: Mean (Standard Deviation); unit: Change in Distance Walked in Meters
Arm/Group | Pirfenidone (2403 mg/d) | Placebo
Number analyzed (Participants) | 171 | 173
Change in Distance Walked in Meters | -45 (140) | -77 (128)

5. Secondary Outcome: Change in Worst Oxygen Saturation by Pulse Oximetry (SpO2) Measurement Observed During the 6-Minute Walk Test
Description: The change from baseline to week 72 in worst oxygen saturation during the 6-Minute Walk Test as measure by Pulse Oximetry (SpO2) Level. It is calculated as the simple difference between baseline SpO2 measurements and week 72 SpO2 measurements.
Time Frame: Baseline to Week 72
Population: A modified intent-to-treat population of all randomized patients who received any amount of study drug is used as the primary population for efficacy and safety analyses. Missing data were imputed by the SSD method if the patient was alive and imputed to 83% if the patient died before the protocol-specified time point.
Measure: Mean (Standard Deviation); unit: Change,Worst Oxygen Saturation (Percent)
Arm/Group | Pirfenidone (2403 mg/d) | Placebo
Number analyzed (Participants) | 171 | 173
Change,Worst Oxygen Saturation (Percent) | -1.9 (3.83) | -1.3 (6.63)

6. Secondary Outcome: Change in Percent Predicted Hemoglobin (Hb)-Corrected Carbon Monoxide Diffusing Capacity (DLco) of the Lungs
Description: The change from baseline to week 72 in Percent Predicted Hemoglobin (Hb)-Corrected Carbon Monoxide Diffusing Capacity (DLco) of the Lungs. It is calculated as the simple difference between baseline DLco measurements and week 72 DLco measurements.
Time Frame: Baseline to Week 72
Population: A modified intent-to-treat population of all randomized patients who received any amount of study drug is used as the primary population for efficacy and safety analyses. Missing data were imputed by the SSD method if the patient was alive and imputed to 0% if the patient died before the protocol-specified time point.
Measure: Mean (Standard Deviation); unit: Change in Percent Predicted DLco
Arm/Group | Pirfenidone (2403 mg/d) | Placebo
Number analyzed (Participants) | 171 | 173
Change in Percent Predicted DLco | -9.8 (12.61) | -9.2 (13.24)

7. Secondary Outcome: Change in Dyspnea Score
Description: The mean change from baseline to week 72 in Dyspnea score was measured by the University of San Diego Shortness of Breath Questionnaire (UCSD SOBQ). The SOBQ is used to assess shortness of breath with various activities of daily living (for example, brushing ones teeth or mowing the lawn). Patients rated the severity of their shortness of breath experienced on an average day during the past week on a 6 point scale (0 to 5),with 0= not at all breathless, 4= severely breathless and 5= Maximally or unable to do because of breathlessness.
Time Frame: Baseline to Week 72
Population: A modified intent-to-treat population of all randomized patients who received any amount of study drug is used as the primary population for efficacy and safety analyses.
  Missing data were imputed by the SSD method if the patient was alive and imputed to a score of 120 if the patient died before the protocol-specified time point.
Measure: Mean (Standard Deviation); unit: Change in Dyspnea Score
Arm/Group | Pirfenidone (2403 mg/d) | Placebo
Number analyzed (Participants) | 171 | 173
Change in Dyspnea Score | 11.9 (24.72) | 13.9 (27.89)

8. Secondary Outcome: Worsening of IPF
Description: Worsening of IPF was defined by the occurrence of any of the following events:
  Acute IPF exacerbation, IPF-related death, Lung transplantation, or Respiratory hospitalization.
Time Frame: Time to acute IPF exacerbation, IPF-related death, lung transplant or respiratory hospitalization, whichever comes first.
Population: as for outcome 3
Measure: Number; unit: Number of Patients Who Worsened
Arm/Group | Pirfenidone (2403 mg/d) | Placebo
Number analyzed (Participants) | 171 | 173
Number of Patients Who Worsened
  Woresening IPF | 24 | 32
  Acute IPF exacerbation | 2 | 1
  IPF-related death | 3 | 6
  Lung transplantation | 2 | 2
  Respiratory hospitalization | 17 | 23
  Patients Censored | 146 | 141

ADVERSE EVENTS:
Arm/Group | Pirfenidone (2403 mg/d) | Placebo
Serious Adverse Events (participants affected / at risk) | 53/171 | 51/173
Other Adverse Events (participants affected / at risk) | 169/171 | 170/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone (2403 mg/d) (N=171) | Placebo (N=173)
Angina Pectoris (Cardiac disorders) | 1 | 1
Angina Unstable (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1
Coronary Artery Disease (Cardiac disorders) | 6 | 0
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 2 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Diverticular Perforation (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Multi Organ Failure (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 5
Bronchitis Viral (Infections and infestations) | 1 | 0
Cholecystitis Infective (Infections and infestations) | 1 | 0
Chronic Sinusitis (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 7 | 7
Pneumonia (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Viral Infection (Infections and infestations) | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Endotracheal Intubation Complication (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 2 | 0
Pelvic Fracture (Metabolism and nutrition disorders) | 1 | 0
Psychosis Postoperative (Injury, poisoning and procedural complications) | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 1
Liver Function Test Abnormal (Investigations) | 2 | 0
Weight Decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastastic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Apraxia (Nervous system disorders) | 0 | 1
Carotid Artery Stenosis (Nervous system disorders) | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Bladder Neck Obstruction (Renal and urinary disorders) | 1 | 0
Glomerulonephritis Rapidly Progressive (Renal and urinary disorders) | 0 | 1
Mesangioproliferative Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 2
Benign Prostatic Hyperpasia (Reproductive system and breast disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 13 | 17
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Aortic Aneurysm (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 2 | 1
Malignant Hypertension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone (2403 mg/d) (N=171) | Placebo (N=173)
Anorexia (Metabolism and nutrition disorders) | 18 | 6
Anxiety (Psychiatric disorders) | 6 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 21 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 54
Decreased appetite (Metabolism and nutrition disorders) | 13 | 9
Depression (Psychiatric disorders) | 10 | 7
Dizziness (Nervous system disorders) | 30 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 34
Headache (Nervous system disorders) | 28 | 25
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 31 | 40
Insomnia (Psychiatric disorders) | 12 | 11
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 6 | 9
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 11 | 11
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 17 | 4
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 7 | 12
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 8
Rash (Skin and subcutaneous tissue disorders) | 58 | 22
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other